CLINICAL TRIAL: NCT02639325
Title: Tumor Related Epilepsy
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160041; 16-N-0041
Record Dates: First submitted 2015-12-23; First posted 2015-12-24 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01-06

CONDITIONS: Epilepsy; Cancer; Brain Neoplasm
Keywords: Brain Tumor; Brain Cancer; Seizure Disorder; Seizures; Natural History
MeSH Terms: conditions — Epilepsy; Neoplasms; Brain Neoplasms; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients who have solitary primary or recurrent brain tumor with associated seizures.

SUMMARY:
Background:

Some people with brain tumors have seizures related to the tumor. This is called tumor-related epilepsy. Usually brain tumors are treated by removing as much of the brain tumor as possible without causing problems. Researchers think this may improve the outcome for people with brain tumors. It may completely relieve or greatly reduce the number of seizures they have.

Objectives:

To evaluate people with brain tumors that are associated with seizures and to offer surgical treatment. Also, to study how surgery affects seizures.

Eligibility:

People age 8 and older who have a brain tumor with associated seizures. They must be willing to have brain surgery to treat their epilepsy.

Design:

Participants will be screened with a review of their medical records.

Participants will have a medical history and physical exam.

Participants will be admitted to the hospital at NIH. They will have

Medical history

Physical exam

Neurological exam

Tests of memory, attention, and thinking

Questions about their symptoms and quality of life

Blood drawn

They may also have:

MRI or CT scan. They will lie on a table that slides in and out of a machine that takes pictures. For part of the MRI, they will get a dye through an intravenous (IV) catheter.

Video electroencephalography monitoring. Electrodes will be placed on the scalp. The participant s brain waves will be recorded while doing normal activities. Participants will be videotaped.

Participants will keep a seizure diary before and after surgery.

Participants will have surgery to remove their brain tumor and the brain area where their seizures start.

They will stay in the hospital up to a week after surgery.

Participants have for follow-up visits at NIH.

DETAILED DESCRIPTION:
Objective

This protocol is being performed to 1) study the natural history and disease pathogenesis in patients with tumor related epilepsy, 2) collect prospective data on seizure outcomes following standard surgical treatment of brain tumors with associated seizures2, 3) follow the clinical course of patients after surgical resection of brain tumors with associated seizures, such as outcomes in seizure activity as they relate to type of tumor and extent of resection, 4) investigate neuropsychological and cognitive outcomes as they relate to surgical and seizure outcomes, 5) evaluate patient reported outcomes such as symptom burden changes as a result of surgical resection in patients with tumor-related epilepsy, 6) examine changes in structural and, when available, functional imaging in the context of tumor related epilepsy before and after surgical resection, 8) investigate molecular markers of tumor-related seizures in tumor and peritumoral specimens and, when available, to compare them to electrophysiological markers of tumor-related seizure activity.

Study Population

Patients 8 years and older with brain tumors and associated seizures may participate in this study.

Study Design

Patients will be screened by study neurosurgeon or neuro-oncologists to verify their confirmed or likely diagnosis of brain tumor and associated seizures. Patients confirmed to have a brain tumor with associated seizures will be offered standard diagnostic and surgical procedures. Non-invasive diagnostic procedures include structural MRI and neuropsychological, cognitive, and outcome assessments which may be performed under other NIH protocols. Some patients may receive functional MRI when clinically indicated, which will be performed under separate NIH protocols. Prior to tumor resection, diagnostic invasive monitoring with intracranial electrodes for further localization of seizure focus and identification of eloquent cortex may be clinically required. In these cases, invasive monitoring will be performed under a separate protocol, 11-N-0051 Epilepsy Surgery. Patients will be followed for three-six months after the surgical procedure to collect prospective data on seizure outcomes following standard surgical treatment of brain

tumors with associated seizures. Patients may also be seen at one year following surgery if medically stable and healthy. Participants in this protocol will not forego other standard treatments for their brain tumor, including chemotherapy and radiation treatment. Participation in this protocol will not preclude eligibility or participation in other NIH clinical trials.

Outcome Measures

The primary outcome measure is the change in seizure frequency, as measured by the Engel scale before and 3-6 months after treatment. Secondary outcome measures include 1) mean Engel Class and absolute and relative change in seizure frequency three-six months after surgery stratified by the type of brain tumor and location and Engel scale, seizure frequency, and mean Engel Class and absolute and relative change in seizure frequency one year after surgery stratified by the type of brain tumor and location; 2) extent of tumor and peri-tumoral resection as seen on MRI imaging and correlation with seizure outcome; 3) changes in neuropsychological and cognitive assessment following surgical resection stratified by location and type of tumor and extent of resection; 4) longitudinal changes in symptom burden and interference scores using established instruments in brain tumor patients; 5) changes in structural imaging following surgical resection; 6) change in the use of anti-epileptic medication; and 7) percentage of patients with permanent neurological side-effects from surgical treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, a candidate must meet all the following criteria:

* Be 8 years of age or older.
* Have solitary primary or recurrent brain tumor with associated seizures. Brain tumor may be diagnosed radiologically. Associated seizures are defined as those with activity starting within three months of radiologic diagnosis of the primary or recurrent tumor. In cases when the timing of seizure activity is unclear with respect to the timing of diagnosis, seizures will be considered associated with the tumor if seizure semiology is consistent with that location. Ongoing seizures are not required. Patients can be included if they have had a single previous seizure. Patients who have not experienced seizures after institution of anti-convulsant therapy are not excluded.

EXCLUSION CRITERIA:

Candidates will be excluded if they:

-At the time of enrollment, lack consent capacity due to cognitive impairment that would make them incapable of understanding the explanation of the procedures in this study. Cognitive capacity to consent will be determined at the time of enrollment. Patients with mental disorders or those patients who are cognitively impaired yet still retain consent capacity will not be excluded. Children may be enrolled if there is a parent or guardian able to consent on their behalf.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One hundred patients, male and female, age 8 or older, with tumor related epilepsy will be enrolled. Patients who withdraw from the protocol will be replaced. The target number of patients completing this study is 100.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-26 (Actual); Primary Completion 2032-07-01 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
change in seizure frequency, as measured by the Engel scale | 3-6 months after surgery
  The primary outcome measure is the Engel scale of patients 3-6 months after treatment. Engel s classification: Class I: patients who were completely seizure free, had auras only, or had convulsions with drug withdrawal only; Class II: rare disabling seizures or nocturnal seizures only; Class III: worthwhile improvement (frequent seizures but fewer than previously); Class IV: no improvement (frequent seizures with unchanged frequency compared to before surgery). Seizure frequency before and after surgical resection will be documented to determine Engel classification.

SECONDARY OUTCOMES:
Mean Engel Class stratified by the type of brain tumor and location | 3-6 months after surgery
  Mean Engel Class three to six months after surgery stratified by the type of brain tumor and location and Engel scale, seizure frequency, and mean Engel Class one year after surgery stratified by the type of brain tumor and location
Extent of tumor and peri-tumoral resection as seen on MRI imaging and correlation with seizure outcome | 3-6 months after surgery
  Extent of tumor resection as seen on MRI imaging and correlation with seizure outcome
Changes in neuropsychological and cognitive assessment following surgical resection stratified by location and type of tumor and extent of resection | 3-6 months after surgery
  Changes in neuropsychological and cognitive assessment following surgical resection stratified by location and type of tumor and extent of resection
Longitudinal changes in symptom burden and interference scores using established instruments in brain tumor patients | 3-6 months after surgery
  Changes in symptom burden and interference with daily activities and quality of life
Changes in structural imaging following surgical resection | 3-6 months after surgery
  Changes in structural imaging following surgical resection
Change in the use of anti-epileptic medication | 3-6 months after surgery
  Percentage of patients who are able to be completely withdrawn from anti-epileptic medication
Percentage of patients with permanent neurological side-effects from surgical treatment | 3-6 months after surgery
  Percentage of patients with permanent neurological side-effects from surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kareem A Zaghloul, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. We will share all IPD that results in a publication on a public repository, as required by most journals. The data will be de-identified and anonymized.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-N-0041.html